CLINICAL TRIAL: NCT04399057
Title: a New Approach: the Use of Shear Wave Elastosonography of the Corpora Cavernosa for the Diagnosis of Erectile Dysfunction.
Brief Title: Shear Wave Elastography New Ultrasound Approach for the Erectile Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Elisabetta Costantini, Chief U.O.C. Chirurgia Urologica ad indirizzo andrologico ed Uroginecologico, University Of Perugia
Other Study IDs: EDSWE1
Record Dates: First submitted 2020-05-12; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Erectile Dysfunction; Penile Diseases
Keywords: erectile dysfunction; elastosonography; penile diseases; International index of erectile function; erectile hardness score
MeSH Terms: conditions — Erectile Dysfunction; Penile Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- andrological patients: shear wave elastosonography of the corpora cavernosa was performed to all patients who went to our clinic for andrological problems. in addition, the International Index of Erectile Function short form (IIEF5) questionnaire and the Erectile Hardness Score (EHS) questionnaire were administered.
  Interventions: Diagnostic Test: shear Wave Elastosonography

INTERVENTIONS:
Diagnostic Test: shear Wave Elastosonography — both the left cavernous body and the right cavernous body are ideally divided longitudinally into three sections: proximal, middle and distal. subsequently for each section of the corpora cavernosa the stiffness of the tissue is calculated by means of a specific Region Of Interest (ROI). the result is expressed in Kilopascals and in a color scale. when registering the stiffness the patient is asked to hold their breath.

SUMMARY:
the study proposes the use of a new non-invasive ultrasound method for the diagnosis of erectile dysfunction. in particular, the shear Wave elastosonosgraphy of the corpora cavernosa will be used. this last method quantitatively measures the rigidity of the analyzed tissues.

DETAILED DESCRIPTION:
erectile function is a complex mechanism in which the elasticity of the tissues that make up the corpora cavernosa is fundamental. indeed, anatomopathological studies have shown that in patients with erectile dysfunction the elastic fibers are replaced by inextensible collagen. the aim of the study is the correlation between penile stiffness measured with this new non-invasive diagnostic method - elastosonography of the corpora cavernosa - and the correlation with validated questionnaires. the international Index of Erectile Function (IIEF5) short form and the erectile Hardness Score (EHS) will be used.

ELIGIBILITY:
Inclusion Criteria:

male who came attended our general andrology clinic between January 2019 to January 2020.

Exclusion Criteria:

1. with: age >80 years or <18 years. , 2
2. diabetes,
3. spinal trauma,
4. treatment with continuous PDE5i,
5. ischemic heart disease for less than 6 months,
6. pelvic surgery for within less than 1 year,
7. hypotestosteronemia (<8 nmol/L),
8. La Peyronie's disease.
9. penile trauma.

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: the population chosen is male, who goes to the clinics for andrological problems.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Shear Wave elastosonografy and Erectile tissues Stiffness. | 15 days
  use of shear wave elastosonography for the diagnosis of erectile dysfunction by measuring the stiffness of the erectile tissue. the rigidity of the cavernous bodies is expressed in numerical values obtained in Kilopascals.
Shear Wave Elastosonography and IIEF5 questionnaire | 15 days
  comparison between the score in the International index of Erectile Function short form questionnaire (minimum value is 5 and maximum value is 25) and the stiffness values obtained by elastosonography with numerical absolute values obtained in kilopascals
Shear Wave elastosonography and EHS questionnaire | 15 days
  comparison between the score in the Erectile hardness Score questionnaire (minimum value is 0 an maximum value is 4) and the stiffness absolute values obtained by elastosonography with the numerical values obtained in kilopascals

SECONDARY OUTCOMES:
cut-off value at elastosonography and erectile dysfunction | 15 days
  The secondary objective aim of the our study is was to establish a cut-off value expressed in kilopascal to the elastosonographic Shear Wave Eelastosonography examination identifies the patient may develop erectile dysfunction due to cavernous tissue rigidity.

CONTACTS AND LOCATIONS:
Locations (1):
- Elisabetta Costantini, Terni, Italy

IPD SHARING:
Plan to Share IPD: No